CLINICAL TRIAL: NCT07168772
Title: The Effect of a Probiotic Administration as an add-on Treatment in Multiple Sclerosis: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: The Effect of a Probiotic Administration as an add-on Treatment in Multiple Sclerosis
Acronym: PROBiMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROBiMS
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactibane Iki (Experimental)
  Interventions: Dietary Supplement: Lactibane Iki
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactibane Iki — Patients will receive a probiotic sachet twice a day for six months. The probiotic, Lactibiane iki (Pileje; Paris, France), is composed of Bifidobacterium lactis LA 304, Lactobacillus acidophilus LA 201, and Lactobacillus salivarius LA 302 and contains 4x10E10 CFU/sachet.
  Arms: Lactibane Iki
Other: Placebo — Patients will receive a placebo (starch) sachet twice a day for six months.
  Arms: Placebo

SUMMARY:
It is a randomized, double-blind, placebo-controlled clinical trial whose general objective of this study is to determine the effects of probiotic administration in multiple sclerosis patients.

80 patients with relapsing-remitting multiple sclerosis will be enrolled in the study. Patients will be randomly assigned to receive either a probiotic (n=40) or a placebo (n=40) stratified by type of medication, gender and use of hormonal contraceptive treatment. They will receive a probiotic (Lactibane Iki) or placebo sachet twice a day for six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-55 years, inclusive
* Diagnosis of RRMS (McDonald Criteria 2017 and Lublin phenotype classification 2014)
* Expanded disability status scale (EDSS) score less than or equal to 5.5
* Patients receiving a first line treatment with teriflunomide or dimethyl fumarate at a stable dose, for at least 24 weeks, or patients who are not receiving treatment because they do not want to receive a DMT after the investigator has informed them of their possible respective benefits and possible adverse events
* At enrollment, the patient is not expected to require a change in DMT
* Patients showing a maximum of two new lesions on MRI prior to inclusion
* Females of childbearing potential must have a negative urine pregnancy test result prior to initiation of study product
* For females of childbearing potential: agreement to use adequate contraceptive methods during the treatment period
* Ability to comply with the study protocol
* Patients must sign and date a written informed consent prior to entering the study

Exclusion Criteria:

* Relapse the month before enrollment
* Presence of a new lesion, indicative of radiological activity, on the MRI performed before starting the study
* Use of corticosteroids the month before enrollment
* Use of antibiotics three months before enrollment
* Taking other forms of symbiotic, probiotic, prebiotic and postbiotic supplements three months before enrollment
* Patients suffering from any type of bowel disease
* Pregnant or breastfeeding or intending to become pregnant during the study.
* Be menopausal
* Be a smoker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in the percentage of Treg cells | 6 months

SECONDARY OUTCOMES:
Immunological profile (percentage of positive cells): Th1 cells; Th17cells; Breg cells; DCs | 6 months
  Immunological profile studied by flow cytometry (percentage of positive cells): Th1 cells; Th17cells; Breg cells; DCs.
Serum levels of NfL, GFAP, cytokines and CRP | 6 months
  Serum levels of NfL and GFAP quantified using a commercially available ultra-sensitive single molecule enzyme-linked immunoarray (SIMOA, Quanterix).
Serum and fecal levels of SCFAs | 6 months
  Serum and fecal levels of SCFAs analyzed using a liquid chromatography tandem mass spectrometry (LC-MS/MS) system.
Microbiota composition analysis | 6 months
  Bioinformatic analysis of the microbiome by the analysis of the total DNA extraction and sequencing of fecal samples and negative control sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Esclerosi Mútiple de Catalunya (Cemcat), Barcelona, Barcelona, Spain